CLINICAL TRIAL: NCT01024010
Title: Phase II Trial of Pentostatin, Cyclophosphamide, and Ofatumumab for Previously Untreated Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL)
Brief Title: Ofatumumab, Pentostatin, and Cyclophosphamide in Treating Patients With Untreated Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC0983; NCI-2009-01437 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC0983 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Results first posted 2018-09-18 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2017-09

CONDITIONS: Chronic Lymphocytic Leukemia; Stage 0 Chronic Lymphocytic Leukemia; Stage I Chronic Lymphocytic Leukemia; Stage I Small Lymphocytic Lymphoma; Stage II Chronic Lymphocytic Leukemia; Stage II Small Lymphocytic Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Small Lymphocytic Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cyclophosphamide; ofatumumab; Pentostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (PCO, closed to accrual as of 8/23/2011) (Experimental): Patients receive induction therapy comprising ofatumumab IV on day 1 (days 1-2 of course 1 only), pentostatin IV over 30 minutes on day 1, and cyclophosphamide IV over 30 minutes on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis; Biological: Ofatumumab; Drug: Pentostatin
- Arm B (PCO with ofatumumab consolidation) (Experimental): Patients receive induction therapy as in Arm A. Patients then receive consolidation therapy comprising ofatumumab IV on day 1. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis; Biological: Ofatumumab; Drug: Pentostatin

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Ofatumumab — Given IV
  Other Names: Arzerra; GSK1841157; HuMax-CD20; HuMax-CD20, 2F2
Drug: Pentostatin — Given IV
  Other Names: (R)-3-(2-Deoxy-.beta.-D-erythro-pentofuranosyl)-3,6,7, 8-tetrahydroimidazo[4,5-d][1,3]diazepin-8-ol; 2'-Deoxycoformycin; CI-825; Co-Vidarabine; Covidarabine; DCF; Deoxycoformycin; Nipent; PD-81565; Pentostatine

SUMMARY:
This phase II trial studies how well giving ofatumumab together with pentostatin and cyclophosphamide works in treating patients with untreated chronic lymphocytic leukemia or small lymphocytic lymphoma. Monoclonal antibodies, such as ofatumumab, can block the ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as pentostatin and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ofatumumab together with pentostatin and cyclophosphamide may be a better way to block cancer growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Arm A: To assess the rate of complete response using pentostatin, cyclophosphamide, and ofatumumab in patients with previously untreated chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) requiring therapy.

II. Arm B: To assess the treatment-free survival rate at 18 months using pentostatin, cyclophosphamide, and ofatumumab induction therapy followed by ofatumumab consolidation in patients with previously untreated CLL or SLL requiring therapy.

SECONDARY OBJECTIVES:

I. Arm A and Arm B: To assess the rate of overall response in patients with previously untreated CLL or SLL requiring therapy and to determine the proportion of patients who achieve a minimal residual disease (MRD) negative state as assessed by flow cytometry in each arm independently.

II. Arm A and Arm B: To monitor and assess toxicity in patients with previously untreated CLL or SLL in each arm independently.

III. Arm A and Arm B: To determine the progression-free survival, treatment-free survival, and duration of response in each arm independently.

IV. Arm A and Arm B: To determine if molecular prognostic parameters (zeta-chain-associated protein [ZAP]-70, cluster of differentiation [CD]38, cytogenetic abnormalities identified by fluorescence in situ hybridization [FISH], immunoglobulin heavy-chain variable-region [IgVH] mutation status, etc) relate to response to therapy in each arm independently.

V. Arm B: To assess the rate of complete response using pentostatin, cyclophosphamide, and ofatumumab induction followed by ofatumumab consolidation in patients with previously untreated CLL or SLL requiring therapy.

VI. Arm B: To evaluate whether consolidation therapy with ofatumumab after pentostatin, cyclophosphamide, and ofatumumab (PCO) induction improves the depth of response.

TERTIARY OBJECTIVES:

I. Arm A and Arm B: To assess the complete and overall response as well as treatment free survival in each arm as compared to a historic control of patients treated with pentostatin, cyclophosphamide, and rituximab in an exploratory manner.

II. Arm A and Arm B: To assess the complete and overall response as well as treatment free survival of patients treated with PCO induction followed by ofatumumab consolidation (Arm B) as compared to patients treated with PCO induction who did not receive ofatumumab consolidation (Arm A) in an exploratory manner.

III. Arm A and Arm B: Assess the mechanisms of ofatumumab induced cell death and explore methods to enhance ofatumumab cytotoxicity.

OUTLINE: Patients are assigned to 1 of 2 treatment arms.

ARM A (closed to accrual as of 8/23/2011): Patients receive induction therapy comprising ofatumumab intravenously (IV) on day 1 (days 1-2 of course 1 only), pentostatin IV over 30 minutes on day 1, and cyclophosphamide IV over 30 minutes on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive induction therapy as in Arm A. Patients then receive consolidation therapy comprising ofatumumab IV on day 1. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 90 days for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL according to the National Cancer Institute (NCI) criteria or SLL according to the World Health Organization (WHO) criteria, including previous documentation of:
* Biopsy-proven SLL
* Diagnosis of CLL according to NCI working group criteria as evidenced by all of the following:

  * Peripheral blood lymphocyte count of > 5,000/mm^3 consisting of small to moderate size lymphocytes, with < 55% prolymphocytes
  * Immunophenotyping consistent with CLL defined as:

    * The predominant population of lymphocytes share both B-cell antigens (CD19, CD20 [typically dim expression], or CD23) as well as CD5 in the absence of other pan-T-cell markers (CD3, CD2, etc.)
    * Clonality as evidenced by kappa or lambda light chain expression (typically dim immunoglobulin expression)
    * Note: splenomegaly, hepatomegaly, or lymphadenopathy are not required for the diagnosis of CLL
  * Before diagnosing CLL or SLL, mantle cell lymphoma must be excluded by demonstrating a negative FISH analysis for t(11;14)(immunoglobulin heavy [IgH]/cyclin D1 [CCND1]) on peripheral blood or tissue biopsy or negative immunohistochemical stains for CCND1 on involved tissue biopsy
* Patients must be previously untreated and meet at least one of the following indications for chemotherapy:

  * Evidence of progressive marrow failure as manifested by the development of or worsening anemia (=< 11 g/dl) and/or thrombocytopenia (=< 100,000/mm^3) not due to autoimmune disease
  * Symptomatic or progressive lymphadenopathy, splenomegaly or hepatomegaly
  * One or more of the following disease-related symptoms:

    * Weight loss > 10% within the previous 6 months
    * Extreme fatigue attributed to CLL
    * Fevers > 100.5 degree Fahrenheit for 2 weeks without evidence of infection
    * Drenching night sweats without evidence of infection
  * Progressive lymphocytosis due to CLL with an increase of > 50% over a two-month period or an anticipated doubling time of less than six months

    * Prior chemotherapy or monoclonal antibody based therapy for treatment of CLL will be considered prior therapy; nutraceutical treatments with no established benefit in CLL (such as epigallocatechin gallate [EGCG], found in green tea or other herbal treatments) will not be considered "prior treatment"
    * Marked hypogammaglobulinemia or the development of a monoclonal protein in the absence of any of the above criteria for active disease are not sufficient for protocol therapy
* Serum creatinine =< 1.5 x upper normal levels (UNL)
* Total bilirubin =< 1.5 x UNL unless due to Gilbert's disease; if total bilirubin is > 1.5 x UNL, a direct bilirubin should be performed and must be < 1.5 mg/dL for Gilbert's to be diagnosed
* Aspartate aminotransferase (AST) =< 3.0 x UNL and alanine aminotransferase (ALT) =< 3.0 x UNL (unless due to hemolysis or CLL)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS): 0, 1, or 2
* Willingness to provide blood samples as required
* Able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

* Any of the following comorbid conditions:

  * New York Heart Association Class III or IV heart disease
  * Recent myocardial infarction (< 1 month)
  * Uncontrolled infection
  * Infection with the human immunodeficiency virus (HIV/acquired immunodeficiency syndrome [AIDS])
  * Infection with known chronic, active Hepatitis C
  * Positive serology for hepatitis B (HB) defined as a positive test for HB surface antigen (HBsAg); in addition, if negative for HBsAg but HB core antibody (HBcAb) positive (regardless of HBsAb status), a HB deoxyribonucleic acid (DNA) test will be performed and if positive the subject will be excluded
* Pregnant women
* Nursing women
* Men or women of childbearing potential who are unwilling to employ adequate contraception
* Other active primary malignancy requiring treatment or limiting survival to =< 2 years
* Any radiation therapy =< 4 weeks prior to registration
* Any major surgery =< 4 weeks prior to registration
* Current use of corticosteroids; EXCEPTION: low doses of steroids (< 10 mg of prednisone or equivalent dose of other steroid) used for treatment of non-hematologic medical conditions; Note: previous use of corticosteroids is allowed
* Active hemolytic anemia requiring immunosuppressive therapy or other pharmacologic treatment; patients who have a positive Coombs test but no evidence of hemolysis are NOT excluded from participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2017-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tait Shanafelt, Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Derived] Strati P, Lanasa M, Call TG, Leis JF, Brander DM, LaPlant BR, Pettinger AM, Ding W, Parikh SA, Hanson CA, Chanan-Khan AA, Bowen DA, Conte M, Kay NE, Shanafelt TD. Ofatumumab monotherapy as a consolidation strategy in patients with previously untreated chronic lymphocytic leukaemia: a phase 2 trial. Lancet Haematol. 2016 Sep;3(9):e407-14. doi: 10.1016/S2352-3026(16)30064-3. Epub 2016 Aug 1. PMID 27570087
- [Derived] Baig NA, Taylor RP, Lindorfer MA, Church AK, LaPlant BR, Pettinger AM, Shanafelt TD, Nowakowski GS, Zent CS. Induced resistance to ofatumumab-mediated cell clearance mechanisms, including complement-dependent cytotoxicity, in chronic lymphocytic leukemia. J Immunol. 2014 Feb 15;192(4):1620-9. doi: 10.4049/jimmunol.1302954. Epub 2014 Jan 15. PMID 24431228

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: PCO: Patients receive 300 mg ofatumumab IV on days 1, cycle 1 and 1000 mg ofatumumab IV on day 2 of cycle 1 and on day 1 of cycles 2-6.
  During cycles 1-6, patients also receive 2 mg/m^2 pentostatin IV over 30 minutes on day 1, 600 mg/m^2 cyclophosphamide IV over 30 minutes on day 1, and 6 mg pegfilgrastim subcutaneously on day 2.
- Arm B: PCO +O: Patients receive 300 mg ofatumumab IV on day 1, cycle 1 and 1000 mg ofatumumab IV on day 2 of cycle 1 and on day 1 of cycles 2-6.
  During cycles1-6, patients also receive 2 mg/m^2 pentostatin IV over 30 minutes on day 1, 600 mg/m^2 cyclophosphamide IV over 30 minutes on day 1, and 6 mg pegfilgrastim subcutaneously on day 2.
  For cycles 7-12, patients receive 1000 mg ofatumumab IV on day 1.
Period: Overall Study
Arm/Group | Arm A: PCO | Arm B: PCO +O
Started | 48 | 34
Completed | 48 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm B: PCO +O: Patients receive 300 mg ofatumumab IV on days 1, cycle 1 and 1000 mg ofatumumab IV on day 2 of cycle 1 and on day 1 of cycles 2-6.
  During cycles1-6, patients also receive 2 mg/m^2 pentostatin IV over 30 minutes on day 1, 600 mg/m^2 cyclophosphamide IV over 30 minutes on day 1, and 6 mg pegfilgrastim subcutaneously on day 2.
  For cycles 7-12, patients receive 1000 mg ofatumumab IV on day 1.
- Total: Total of all reporting groups
Arm/Group | Arm A: PCO | Arm B: PCO +O | Total
Number analyzed (Participants) | 48 | 34 | 82
Age, Continuous [Median (Full Range); unit: years] | 65 [50 to 83] | 59 [40 to 79] | 63 [40 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 5 | 19
  Male | 34 | 29 | 63
Region of Enrollment [Number; unit: participants]
  United States | 48 | 34 | 82

OUTCOME MEASURES:

1. Primary Outcome: Arm A: Percentage of Complete Responses
Description: In Arm A: PCO, the primary endpoint of this trial is the percentage of complete responses. The NCI Working Group criteria was used to assess response to therapy:
  A Complete Response (CR) is briefly defines as the absence of lymphadenopathy, no heptomegaly nor splenomegaly, neutrophils greater than 1500/ul, platelets > 100,000/ul, hemoglobin >11.0 gm/dl, and peripheral blood lymphocytes <4000uL.
Time Frame: 7 months
Population: All patients that began Arm A protocol treatment were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: PCO
Number analyzed (Participants) | 48
percentage of participants | 46 [31 to 61]

2. Primary Outcome: Arm B: Treatment-free Survival at 18 Months
Description: The primary endpoint Arm B: PCO+O is treatment-free survival rate at 18 months. An event for treatment-free survival will be defined as initiation of subsequent therapy for CLL or death due to any cause. All patients meeting the eligibility criteria who have signed a consent form and have begun treatment will be evaluable for event-free survival at 18 months. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true success proportion will be calculated.
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: PCO | Arm B: PCO +O
Number analyzed (Participants) | 48 | 34
percentage of participants | 87.5 [74.3 to 94.2] | 94.1 [78.5 to 98.5]

3. Secondary Outcome: Overall Response Rate
Description: The overall response rate will be estimated by the total number of complete or partial responses (CCR, CR, CRi, nPR, or PR) divided by the total number of evaluable patients. Responses will be evaluated using NCI Working Group criteria. Minimum requirements for a Partial Response (PR) requires:
  * 50% decrease in peripheral blood lymphocyte count from the baseline
  * 50% reduction in the sum of the products of the largest measured node or nodal masses on physical examination.
  * 50% reduction in size of liver and/or spleen
  * 50% improvement in neutrophils, platelets and hemoglobin
Time Frame: 14 months
Population: All patients were evaluable for this endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: PCO | Arm B: PCO +O
Number analyzed (Participants) | 48 | 34
percentage of participants | 96 [86 to 99] | 97 [85 to 100]

4. Secondary Outcome: Depth of Response After Ofatumumab Consolidation
Description: The proportion of patients with an improvement in depth of response with the addition of ofatumumab consolidation after PCO induction will be estimated by the number of patients with improvement in response from the time of response evaluation at the completion of PCO to the time of response evaluation at the completion of ofatumumab consolidation divided by the total number of evaluable patients. The hierarchy for depth of response will be in the following increasing order: SD, PR, nPR, CR/CRi with MRD+, CR/CRi with MRD-. An improvement in depth of response will be defined as an improvement of at least one level in the hierarchy. Exact binomial 95% confidence intervals for the true overall improvement rate will be calculated.
Time Frame: 14 months
Population: Thirty-one out of the 34 patients registered to Arm B: PCO+O began consolidation, 28 were evaluated for response at the end of consolidation treatment (3 patients did not return for response evaluation at the end of treatment).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: PCO | Arm B: PCO +O
Number analyzed (Participants) | 0 | 28
percentage of participants |  | 25 [11 to 45]

5. Secondary Outcome: Treatment-free Survival
Description: Treatment-free survial is defined as the time from registration to the date of initiation of subsequent treatment for CLL or death due to any cause. The distribution of treatment-free survival will be estimated using the method of Kaplan-Meier.
Time Frame: up to 5 years from registration
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: PCO | Arm B: PCO +O
Number analyzed (Participants) | 48 | 34
months | 56.6 [50.16 to NA] — There have not been a sufficient number of events to calculate the upper 95% confidence limit. | NA [33.8 to NA] — There have not been a sufficient number of events to calculate the median and upper 95% confidence limit.

ADVERSE EVENTS:
Arm/Group | Arm A: PCO | Arm B: PCO +O
Serious Adverse Events (participants affected / at risk) | 10/48 | 6/34
Other Adverse Events (participants affected / at risk) | 48/48 | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: PCO (N=48) | Arm B: PCO +O (N=34)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Mobitz (type) II atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: PCO (N=48) | Arm B: PCO +O (N=34)
Anemia (Blood and lymphatic system disorders) | 40 (179) | 32 (183)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (2)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 18 (29) | 5 (10)
Vomiting (Gastrointestinal disorders) | 6 (10) | 2 (6)
Chills (General disorders) | 3 (4) | 1 (1)
Fatigue (General disorders) | 13 (25) | 6 (13)
Fever (General disorders) | 13 (16) | 12 (15)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 1 (1) | 3 (3)
Allergic reaction (Immune system disorders) | 0 (0) | 3 (7)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (2)
Anorectal infection (Infections and infestations) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 7 (9) | 8 (12)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Peripheral nerve infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 2 (2) | 2 (2)
Upper respiratory infection (Infections and infestations) | 16 (23) | 19 (40)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 18 (118)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 23 (55) | 26 (96)
Platelet count decreased (Investigations) | 33 (205) | 30 (248)
Weight loss (Investigations) | 2 (2) | 0 (0)
White blood cell decreased (Investigations) | 27 (70) | 28 (150)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 (8) | 4 (4)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 5 (6) | 2 (2)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Lymphedema (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes